CLINICAL TRIAL: NCT03771508
Title: PillCam SB3 Registry for Development and Validation of Improved Algorithms for GI Pathologies Detection
Brief Title: Prospective Collection of PillCam SB3 Videos and Raw Data Files for Future Developments (SODA)
Acronym: SODA
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT18014
Record Dates: First submitted 2018-12-07; First posted 2018-12-11 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-07

CONDITIONS: Small Intestine Disease; Small Intestine Cancer; Small Intestinal Ulcer Bleeding; Small Intestine Obstruction; Small Intestine Adenocarcinoma; Small Intestine Polyp

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

GROUPS / COHORTS (1):
- PillCam SB3 procedure: Subjects with normal/abnormal PillCam SB3 procedure

SUMMARY:
Observational, Multicenter, Post-market, Minimal risk, Prospective data collection of PillCam SB3 videos (including PillCam reports) and raw data files and optional collection of Eneteroscopy reports

DETAILED DESCRIPTION:
Up to 8000 PillCam SB3 videos (including PillCam reports) and raw data files will be collected in up to 50 medical centers in the US. Study duration is up to 7 years from IRB approval.

Medical center study sites will provide relevant videos (including PillCam reports) and raw data from patients who underwent SB3 procedures.

Per patient demographic data will be also collected to provide a description of the study population characteristics and disposition.

Additional Standard of care data collection might be performed (optional). This data will include a de-identified Eneteroscopy report, from patients enrolled to the study and referred to Eneteroscopy procedure (all types of Eneteroscopies), following findings identified during the PillCamTM SB procedure, as part of the standard of care procedure. This data might be collected retrospectively for enrolled patients who underwent an Eneteroscopy procedure. The de-identified reports will be used by MDT GI research and development team to further develop and validated SB capsule localization.

Study subjects will not undergo any additional procedures, nor will their diagnosis and subsequent treatment pathway be changed for the purpose of the registry.

The data will be used by MDT GIs research and development team for the development and validation of improved and new detectors in the PillCam software.

The videos (including PillCam reports) and raw data files will be de-identified at the medical center by representatives who are authorized and delegated to review medical records, prior to providing them to the sponsor. All data in the study- videos, reports, raw data files and demographic information will be de-identified in a manner that is untraceable by the sponsor clinical study team members.

ELIGIBILITY:
Inclusion Criteria:

* All SB3 cases collected during standard of care procedures.
* The subject received an explanation and understands the nature of the study and provided oral consenting

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent Standard of Care SB3 procedure
Sampling Method: Non-Probability Sample
Enrollment: 3712 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Prospective collection of PillCam SB3 videos | Up to 7 years from study approval
  sponsor database will be expanded with images of pathologies and normal mucosa for future development and validation of improved algorithms for GI pathologies detection with the PillCam platform

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Sojourner, Study Director — Medtronic
Locations (30):
- United States (30):
  - Birmingham Gastroenterology Associates, Birmingham, Alabama
  - Gastroenterology & Liver Institute, Escondido, California
  - Amicis Research Center, Valencia, California
  - Medical Research Center of Connecticut, Hamden, Connecticut
  - Encore Borland-Groover, Jacksonville, Florida
  - Research Associates of South Florida, Miami, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - Digestive Healthcare of GA, Atlanta, Georgia
  - The University of Kansas Medical Center, Kansas City, Kansas
  - Capital Digestive Care, Chevy Chase, Maryland
  - Gastro Center of Maryland, Columbia, Maryland
  - Woodholme Gastroenterology Associates, Pikesville, Maryland
  - UMass Memorial Health Care, Worcester, Massachusetts
  - Digestive Health Associates, Farmington Hills, Michigan
  - Clinical Research Professionals, Chesterfield, Missouri
  - The Children's Mercy Hospital, Kansas City, Missouri
  - Atlantic Digestive Health Institute, Morristown, New Jersey
  - Albany Gastroenterology Consultants, Albany, New York
  - Erber M.D. PC, Brooklyn, New York
  - Northwell Health - Cohen Children's Medical Center of New York, Lake Success, New York
  - New York Gastroenterology Associates, New York, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - The Toledo Clinic, Toledo, Ohio
  - Digestive Disease Specialists Inc, Oklahoma City, Oklahoma
  - USDH Clinical Research, Exton, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Palmetto Primary Care, Summerville, South Carolina
  - Austin Gastro, Austin, Texas

IPD SHARING:
Plan to Share IPD: No
Patient data will not be shared.